CLINICAL TRIAL: NCT06807567
Title: Understanding Risk Factors for Progressive Chronic Kidney Disease in Malawi to Inform Interventions for Earlier Detection ad Prevention (Impso Study)
Brief Title: Acceptability and Feasibility of Interventions for Integrated Care of Chronic Kidney Disease With Other Long-term Health Conditions in Malawi: a Qualitative Study
Acronym: Impso
Status: Not yet recruiting | Type: Observational
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Wellcome Trust (Liverpool Clinical PhD Programme) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 24-057
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease(CKD); Multimorbidity; Long-term Health Conditions
Keywords: integrated care; chronic kidney disease; long-term conditions; qualitative research; Malawi
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Policy Making

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients and caregivers: Patients aged 18 years and over with CKD, or at risk of CKD, who have at least one other long-term condition, and who are receiving care at either Queen Elizabeth Central Hospital in Blantyre, Chiradzulu District Hospital, Namadzi or Ndunde primary health care centres. Caregivers will be the caregivers of patients meeting these conditions.
  Interventions: Other: Receipt of healthcare for long-term conditions
- Healthcare workers: Healthcare workers, aged 18 years and over, providing care for patients with CKD and other long-term health conditions at Queen Elizabeth Central Hospital in Blantyre, Chiradzulu District Hospital, Namadzi or Ndunde primary health care centres.
  Interventions: Other: Provision of healthcare
- Policy makers: Policy makers with roles in policy making related to CKD and other long-term health conditions in Malawi.
  Interventions: Other: Policy making

INTERVENTIONS:
Other: Receipt of healthcare for long-term conditions — The patient participants are people who are already receiving healthcare for CKD and/or hypertension, diabetes, HIV, heart failure and/or stroke at one of the named study sites, for at least 6 months prior to recruitment into this qualitative study. The caregiver participants are caregivers for patients meeting these criteria.
  Groups: Patients and caregivers
Other: Provision of healthcare — The healthcare worker participants are all providing care to patients with long-tem conditions, at one of the names study sites
  Groups: Healthcare workers
Other: Policy making — The policy makers recruited to this study will be individuals involved in policy making for long-term conditions in Malawi
  Groups: Policy makers

SUMMARY:
The burden of chronic kidney disease (CKD) is rising globally, but disproportionately impacting on low- and middle-income countries (LMIC) including Malawi, which have the fewest resources to manage it. Furthermore, CKD is the leading cause of catastrophic health expenditure worldwide, largely due to the extremely high costs of kidney replacement therapy (KRT) for people with kidney failure. Access to KRT remains limited in many settings, including Malawi, where there is only one nephrologist for a population of over 21 million. It is therefore essential to diagnose and treat CKD in its early stages, to facilitate earlier and more cost-effective treatment to prevent its progression to advanced disease which is associated with increased risks of kidney failure and of cardiovascular morbidity and mortality. CKD is usually asymptomatic in its early stages, so early diagnosis and treatments requires access to key diagnostic tests, in addition to strategies for channelling resources to those at the highest risk.

The causes of CKD are diverse, particularly in LMIC settings where the increasing prevalence of non-communicable diseases intersects with ongoing high burdens of infectious diseases, malnutrition, and many other social and environmental determinants of kidney health. The World Health Organization recommends integrated approaches to improve equity of quality care for people living with long-term conditions, and CKD would be amenable to integrated approaches, however CKD has been neglected from global NCD agendas and there is little data to guide the most effective methods for integrating its care with other long-term conditions (such as hypertension, diabetes and HIV infection), particularly in low-income settings such as Malawi.

The aim of this study is to explore current experiences of care for CKD and related long-term conditions, and to qualitatively evaluate the acceptability and feasibility of different potential approaches to integrating their care, amongst different stakeholders groups in Malawi.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria for each of the participant groups described above are as follows:

Patients:

1. Adults aged ≥ 18 years
2. Diagnosed with CKD, or at risk of CKD, AND at least one other long-term health condition out of:

   * Hypertension
   * Diabetes mellitus
   * HIV infection
   * Heart failure
   * Stroke (See Table 1 for diagnostic inclusion criteria for each of the above conditions)
3. Receiving outpatient care at one of the selected study sites, for at least 6 months

Caregivers:

1. Adults aged ≥ 18 years
2. Identified by a patient meeting the above inclusion criteria to be their primary caregiver

Healthcare workers:

* Adults aged ≥ 18 years
* Currently employed as a healthcare worker at either QECH, Chiradzulu District Hospital, Ndunde Health Centre or Namadzi Health Centre.
* Working in an outpatient clinic environments where care is delivered for patients with any of the above conditions, which may include (but is not limited to) the following:

  * CKD clinic (QECH)
  * Hypertension clinic (QECH)
  * Diabetes clinic (QECH)
  * HIV clinic (all study locations, including the Lighthouse clinic at QECH)
  * Cardiology /chest clinic (QECH)
  * General non-communicable disease (Chiradzulu District Hospital and its referring primary health centres)

Policy makers

* Adults aged ≥ 18 years
* Identified through stakeholder mapping and/or snowball sampling to have a leading role relevant to planning, managing and implementing services and/or policies for NCDs and/or other LTCs.

Exclusion Criteria:

* • Under 18 years of age

  * Acute physical or mental illness, which requires urgent treatment and might impact on ability to participate in and complete interview
  * Current hospital inpatient
  * Unable to participate in interview due to severe communication difficulties (e.g. aphasia), confusion or behavioural disturbance
  * Declines consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - We will recruit adults aged 18 years and older from the following stakeholder groups:
  * Patients
  * Caregivers
  * Healthcare workers (HCWs)
  * Policy makers
  Patients will be adults with, or at risk of, CKD and at least one other long-term health condition, who receive outpatient care at Queen Elizabeth Central Hospital (QECH) in Blantyre, Chiradzulu District Hospital or primary health centres within Chiradzulu district.
  * Caregivers of patients from meeting eligibility criteria will also be invited to participate, if they are identified by the patient to be their primary caregiver.
  * Healthcare workers (HCWs) will be recruited from amongst staff working at any of the named study locations, whose role involves caring for patients with CKD and/or other long-term health conditions.
  * Policy makers will be individuals with leading roles in planning, managing and implementing services and policies for non-communicable diseases and/or other long-term conditions in Malawi
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-17 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Codes and themes | 6 months from end of data collection
  The outcomes of this study will be the codes and themes identified through thematic analysis of the interview and focus group discussion transcripts.

CONTACTS AND LOCATIONS:
Locations (1):
- Malawi Liverpool Wellcome Clinical Research Programme, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Access may be granted to pseudonymised interview transcripts to approved researchers for the purposes of secondary analyses, only following completion of the analysis and subject to approval by the Malawi Liverpool Wellcome Programme (MLW) research strategy group.
Supporting Information: CSR, Analytic Code
Time Frame: After completion of the main analysis, and up to a maximum of 5 years after completion fo the study
Access Criteria: Subject to application to the MLW research strategy group and their approval